CLINICAL TRIAL: NCT06601530
Title: Investigation of the Efficacy of Transversus Thoracic Muscle Plane Block in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Transversus Thoracic Muscle Plane Block (TTMP) on Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bensu Tavelli, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 367860
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Bypass; Anesthesia, Conduction; Nerve Block; Pain, Postoperative
Keywords: Transversus thoracic muscle plane block, postopertive pain, sternotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Thoracic Muscle Plane Block Group (Experimental): Transversus thoracic muscle plane block is a single-shot nerve block technique that provides analgesia for the anterior chest wall
  Interventions: Procedure: Transversus Thoracic Muscle Plane Block; Drug: Tramadol
- Control Group (Active Comparator)
  Interventions: Drug: Tramadol

INTERVENTIONS:
Procedure: Transversus Thoracic Muscle Plane Block — Transversus thoracic muscle plane block is a single-shot nerve block technique that provides analgesia for the anterior chest wall Tramadol IV PCA (Patient Controlled Analgesia): Basal infusion 0.2 mg/kg/h, bolus 20 mg, lock time 20 minutes
  Other Names: Tramadol
  Arms: Transversus Thoracic Muscle Plane Block Group
Drug: Tramadol — Tramadol IV PCA (Patient Controlled Analgesia): Basal infusion 0.2 mg/kg/h, bolus 20 mg, lock time 20 minutes

SUMMARY:
In this prospective and controlled study, the investigators investigated the effect of transversus thoracic muscle plane block (TTMP) on analgesia in patients who undergo coronary artery bypass graft (CABG) surgery with median sternotomy. For this purpose, the investigators aimed to compare the hemodynamic responses to surgical incision and sternotomy and, pain intensity, total analgesic consumption, additional analgesic requirements of the patients in the first 24 hours after extubation under postoperative patient-controlled analgesia (PCA) adminisration.

DETAILED DESCRIPTION:
Forty-six patients aged 18-70 years, ASA class I-III, who undergo CABG surgery were included in our study. The patients were randomized into the TTKPB group and the control group. Heart rate (HR) and mean arterial pressure (MAP) were recorded before peroperative induction, before skin incision, after skin incision, before sternotomy and after sternotomy. PCA with tramadol was applied after extubation and "Numeric rating scale" NRS scores, total tramadol consumption, number of requests and additional analgesic requirements were recorded at 0, 1, 2, 4, 8, 12 and 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) classification I-III
* Coronary artery bypass graft operation with median sternotomy under elective conditions

Exclusion Criteria:

* Refusing to participate in the study
* Under 18 and over 70
* ASA class IV and above
* EF (Ejection Fraction) < 40%
* Emergency surgery or reoperation
* Intraaortic balloon pump placement
* Known allergy to local anesthetics
* Coagulation disorder
* Infection at the block site
* History of sternotomy
* Those with chronic pain complaints and long-term use of analgesics
* Patients who could not be extubated within 12 hours after the operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) at rest | Postoperative 24 hours
  Numeric Rating Scale (NRS) for postoperative pain
Numeric Rating Scale (NRS) during coughing | Postoperative 24 hours
  Numeric Rating Scale (NRS) for postoperative pain
Mean arterial pressure | Postoperative 24 hours
  Postoperative 0, 1, 2, 4, 8, 12 and 24 hours
Heart rate | Postoperative 24 hours
  Postoperative 0, 1, 2, 4, 8, 12 and 24 hours
Mean arterial pressure | Peroperative
  Peroperative induction, before skin incision, after skin incision, before sternotomy and after sternotomy.
Heart rate | Peroperative
  Peroperative induction, before skin incision, after skin incision, before sternotomy and after sternotomy.
Bispectral Index (BIS) | Peroperative
  Peroperative induction, before skin incision, after skin incision, before sternotomy and after sternotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Lale Yüceyar, Prof, Study Chair — Istanbul University - Cerrahpasa; Nevzat Cem Sayılgan, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF

REFERENCES:
- [Background] Fujii S, Vissa D, Ganapathy S, Johnson M, Zhou J. Transversus Thoracic Muscle Plane Block on a Cadaver With History of Coronary Artery Bypass Grafting. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):535-537. doi: 10.1097/AAP.0000000000000607. No abstract available. PMID 28632672
- [Background] Dogan Baki E, Kavrut Ozturk N, Ayoglu RU, Emmiler M, Karsli B, Uzel H. Effects of Parasternal Block on Acute and Chronic Pain in Patients Undergoing Coronary Artery Surgery. Semin Cardiothorac Vasc Anesth. 2016 Sep;20(3):205-12. doi: 10.1177/1089253215576756. Epub 2015 Apr 21. PMID 25900900
- [Background] Hamed MA, Boules ML, Sobhy MM, Abdelhady MA. The Analgesic Efficacy of Ultrasound-Guided Bilateral Transversus Thoracic Muscle Plane Block After Open-Heart Surgeries: A Randomized Controlled Study. J Pain Res. 2022 Mar 5;15:675-682. doi: 10.2147/JPR.S355231. eCollection 2022. PMID 35281480
- [Background] Shokri H, Ali I, Kasem AA. Evaluation of the Analgesic Efficacy of Bilateral Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Post-Sternotomy Pain: A Randomized Controlled Trial. Local Reg Anesth. 2021 Nov 12;14:145-152. doi: 10.2147/LRA.S338685. eCollection 2021. PMID 34803399
- [Background] Abdelbaser II, Mageed NA. Analgesic efficacy of ultrasound guided bilateral transversus thoracis muscle plane block in pediatric cardiac surgery: a randomized, double-blind, controlled study. J Clin Anesth. 2020 Dec;67:110002. doi: 10.1016/j.jclinane.2020.110002. Epub 2020 Jul 24. PMID 32717448
- [Background] Kaya C, Dost B, Dokmeci O, Yucel SM, Karakaya D. Comparison of Ultrasound-Guided Pecto-intercostal Fascial Block and Transversus Thoracic Muscle Plane Block for Acute Poststernotomy Pain Management After Cardiac Surgery: A Prospective, Randomized, Double-Blind Pilot Study. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt A):2313-2321. doi: 10.1053/j.jvca.2021.09.041. Epub 2021 Oct 1. PMID 34696966
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179